CLINICAL TRIAL: NCT03986632
Title: Tundra Gifts: Harvesting Local And Regional Resources To Prevent Obesity Among Alaska Native Children In Remote, Underserved Communities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Alaska Fairbanks (Other)
Collaborators: Pacific Institute for Research and Evaluation (Other); University of Alaska Anchorage (Other); State of Alaska Department of Health and Social Services (Unknown); Grand Valley State University (Other); Alaska Native Tribal Health Consortium (Other)
Responsible Party: Principal Investigator, Andrea Bersamin, Associate Professor, University of Alaska Fairbanks
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-69001-27544
Record Dates: First submitted 2019-06-02; First posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Childhood Obesity
Keywords: Healthy Eating; Alaska Native; Traditional Foods
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tundra gifts program (Experimental)
  Interventions: Behavioral: Tundra Gifts
- Comparison (No Intervention)

INTERVENTIONS:
Behavioral: Tundra Gifts — Tundra Gifts is a home-focused intervention delivered by community health workers (CHW) that focuses on promoting healthy eating and an active lifestyle among 3-5 year olds through family and community partnerships. Primary caregivers will attend monthly interactive education session, receive a monthly gift basket that includes resources and supplies to support behavior change at home and receive ongoing social support through a Facebook site.
  Arms: Tundra gifts program

SUMMARY:
The long-term goal of this community based participatory research project is to prevent obesity in 3-5 year old Alaska Native children in remote communities.

Investigators will design and evaluate a culturally responsive, home-focused intervention, Tundra Gifts, that links early childhood education programming (i.e. Head Start) and federal food assistance programs (i.e. WIC and SNAP) with primary caregivers to support healthy eating and an active lifestyle using a cluster-randomized design. The intervention integrates behavior change theory with Indigenous traditional knowledge. Primary caregivers will attend monthly interactive education session, receive a monthly gift basket that includes resources and supplies to support behavior change at home and receive ongoing social support through a Facebook site. Investigators will also evaluate key process indicators of Tundra Gifts to understand the impact on outcomes of variations in persons and settings and to enhance the generalizability of findings.

ELIGIBILITY:
Inclusion Criteria:

* 3-5 year old children enrolled in Head Start and their primary caregiver in Yup'ik Alaska Native communities

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in age- and sex-specific BMI percentiles and z-scores | twice annually for 3 years
Change in child intake of vegetables and fruit | twice annually for 3 years
  24-hour recall in combination with a 2-day food record
Change in child intake of vegetables and fruit | twice annually for 3 years
  Skin carotenoid meter using reflection spectroscopy (veggie-meter)
Change in child intake of sugar sweetened beverages | twice annually for 3 years
  Hair biomarker of sugar using N and C stable isotope ratios
Change in child intake of sugar sweetened beverages | twice annually for 3 years
  24-hour recall in combination with a 2-day food record
Change in child screen time | twice annually for 3 years
  Screen time questionnaire
Change in child physical activity | twice annually for 3 years
  Physical activity questionnaire

SECONDARY OUTCOMES:
Change in adult attitudes and beliefs around healthy eating and active lifestyle | twice annually for 3 years
  Attitudes and beliefs questionnaire
Change in adult BMI | twice annually for 3 years
Change in adult intake of vegetables and fruit | twice annually for 3 years
  skin carotenoid meter using reflection spectroscopy (veggie-meter)